CLINICAL TRIAL: NCT06749210
Title: DANCE-BASED AVENUES TO ADVANCE NONPHARMACOLOGIC TREATMENT OF CHEMOTHERAPY EFFECTS (DAANCE): A MULTICENTER TRIAL
Brief Title: DAANCE FOR CHEMOTHERAPY-INDUCED NEUROPATHY
Acronym: DAANCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Yale University (Other); Emory University (Other)
Responsible Party: Principal Investigator, Lise Worthen-Chaudhari, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-24277; R01AG084676 (NIH); OSU-24277 (Other: Ohio State Comprehensive Cancer Center)
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-07

CONDITIONS: Cancer of the Breast; Chemotherapy-induced Neuropathy
Keywords: survivorship; music; dance
MeSH Terms: conditions — Breast Neoplasms | interventions — Aryl Hydrocarbon Receptor Nuclear Translocator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): 4 weeks of usual care followed by optional 1-way crossover to 8 weeks of Intervention (partnered, adapted tango dance)
- Experimental (Experimental): 8 weeks of intervention (partnered, adapted tango dance)
  Interventions: Behavioral: Tango

INTERVENTIONS:
Behavioral: Tango — The intervention being studied is a 16 session intervention (2x4-week modules), delivered over an 8-week period by community-based individuals with expertise in dance and patient care and certified in Adapted Tango or AdapTango dance instruction. Steps available to teach, including order and cues to teach them, are detailed in Hackney's AdapTango manual. All steps are based on the Argentine Tango steps that emerged within working class community centers in Buenos Aires, Argentina (milongas) in the late 1800s and have been adapted by the investigators for use as medical exercise among people with mobility deficits. Of note, Argentine Tango is distinct from, and the precursor for, the American Tango style of competitive ballroom dance: where American Tango highlights showmanship and complicated footwork, Argentine Tango prioritizes connection between partners and musicality within a basic walk motion.
  Arms: Experimental

SUMMARY:
Up to 80% of breast cancer survivors experience chemotherapy-induced neuropathy that impairs quality of life and increases fall risk long into survivorship, yet treatment options for neuropathy remain limited. The successful treatment will target neurophysiologic mechanisms for restoring function while addressing patient-reported symptoms and participation in treatment. Toward this end, the investigators propose to study a noninvasive, social sensorimotor intervention - Adapted Argentine Tango - which targets motor control restoration, symptom alleviation, and treatment participation in concert.

DETAILED DESCRIPTION:
This study will investigate a noninvasive, social, sensorimotor intervention which targets motor control restoration, symptom alleviation, and treatment participation in concert: partnered Adapted Argentine Tango (Tango). This project will expand the investigators' pilot work (R21-AG068831) into a multicenter clinical trial designed to investigate the effect of social dance on sensory relief, functional restoration, and key mechanisms of action among a diverse cohort of BC survivors suffering from chronic chemotherapy-induced sensorimotor deficits.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer (BC) diagnosis of Stage I-IV including metastatic disease
* completed taxane-based chemotherapy for BC at least 3 months ago (no limit on how long ago)
* symptomatic for chemotherapy-induced neuropathy (self-report)
* postural control score that indicates potential fall-risk
* able to understand and comply with directions associated with testing and study treatments

Exclusion Criteria:

* pre-existing vestibular dysfunction
* poorly controlled diabetes (hgA1C>=8)
* non-ambulatory (assistive and prosthetic devices allowed)
* hearing impairment resulting in less than 10% hearing bilaterally
* contraindication to participate in the experimental physical activity per the treating oncologist due to additional condition (e.g., herniated disc, unstable bone metastases)
* currently in activity-based therapy (e.g., physical therapy, occupational therapy). May enroll if still meet eligibility criteria once activity-based therapy is complete.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2029-08-15 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcome (PRO) - CIN sensation | 4 weeks
  Sensation of numbness/tingling on 0-10 scale; minimum value 0 (no numbness/tingling); maximum value 10 (worst numbness/tingling)
Dual-task function | 4 weeks
  Ability to move and think at the same time as measured by time to complete the Timed-Up-and-Go (TUG) test with concurrent cognitive task (i.e., counting backward by some number while completing a defined movement task)

SECONDARY OUTCOMES:
Patient-Reported Outcome (PRO) - hot/cold sensation | 4 weeks; 8 weeks; 12 weeks
  Sensation of hot and/or cold (11 point Likert scale).
EORTC-CIPN 20 | mid-intervention (4weeks); post -intervention (8 weeks); 1 month follow up post intervention
  European Organization for Research and Treatment of Cancer Chemotherapy-Induced Peripheral Neuropathy symptoms inventory (CIPN 20),
Brief Fatigue Inventory | 4 weeks; 8 weeks; 12 weeks
  The Brief Fatigue Inventory (BFI) is a short questionnaire used to quickly assess the severity of fatigue, particularly in cancer patients, by measuring both the level of tiredness and how much fatigue interferes with daily activities, allowing for rapid evaluation in clinical settings or research studies; it consists of nine items where patients rate their fatigue on a scale from 0 to 10, with higher scores indicating greater fatigue severity.
Brief Pain Inventory | 4 weeks; 8 weeks; 12 weeks
  The Brief Pain Inventory (BPI) is a self-reported questionnaire used to assess the severity of pain and how much it interferes with a person's daily activities, including aspects like mood, work, sleep, and social interactions. It measures pain intensity on a scale from 0 (no pain) to 10 (worst pain imaginable) across different timeframes (current, average, worst pain) while also evaluating the impact of pain on various life functions on a similar 0-10 scale; it comes in both short and long forms, with the long form including more detailed questions about pain characteristics and treatment history.
Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | 4 weeks; 8 weeks; 12 weeks
  The PRO-CTCAE assessment, which stands for "Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events," is a measurement system designed by the National Cancer Institute (NCI) to capture and evaluate the symptomatic side effects experienced by cancer patients during clinical trials, allowing patients to self-report on the frequency, severity, interference, and presence/absence of symptoms like pain, fatigue, nausea, and skin reactions, providing a more patient-centric perspective on treatment toxicity compared to clinician-based assessments alone.
Physical Health Questionnaire-2 (PHQ-2) | 4 weeks; 8 weeks; 12 weeks
  The PHQ-2 asks how often a patient has experienced depressed mood or anhedonia in the last two weeks
Generalized Anxiety Questionnaire | 4 weeks; 8 weeks; 12 weeks
  Each question has a 4-point scale, ranging from 1, "not at all", to 4, "nearly every day".
Falls | 4 weeks; 8 weeks; 12 weeks; 6 months following intervention end
  Report of whether you have fallen or lost your balanced since we last spoke with you
The Mini Balance Evaluation Systems Test (MiniBEST) | 4 weeks (Control group); 8 weeks (Intervention group)
  The Mini-BESTest (Balance Evaluation Systems Test) is a 14-item test that measures balance, functional mobility, and gait by assessing dynamic balance, anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait.
Biomechanical measures of postural control | 4 weeks; 8 weeks; 12 weeks
  Postural sway while standing still with eyes closed.
Six minute walk test (6mwt) | 4 weeks; 8 weeks
  A "6 minute walk test" (6MWT) is a medical assessment where a person walks as far as they can in a designated area for six minutes, with the primary goal of measuring their functional exercise capacity, usually used to evaluate patients with conditions affecting their breathing or mobility, like heart failure or lung disease; the distance walked during those six minutes is the key measurement recorded as the "6-minute walk distance" (6MWD)
Gait stability | 4 weeks; 8 weeks
  Stability between gait strides over the period of the 6mwt.
Upper Extremity Function | 4 weeks; 8 weeks; 12 weeks
  We assess upper extremity function using the "back scratch test" which measures upper body flexibility and shoulder mobility. Participants reach both hands toward each other behind their backs and staff measure the distance remaining between their fingertips.

OTHER OUTCOMES:
Brain Activity | 4 weeks (Control group); 8 weeks (Intervention group)
  Electroencephalography (EEG)-based measures of brain activity during performance of functional activities (e.g., walking standing, thinking). We will analyze Alpha and Gamma frequencies with regard to amplitude and timing of peak activity.
Blood-based biomarkers of inflammation | 4 weeks (Control group); 8 weeks (Intervention group)
  IL-6, IL-7, IL-8, IL-9, IL-10, TNF-alpha, IRN-gamma, MCP-1
Blood-based biomarkers of neurotoxity | 4 weeks (Control group); 8 weeks (Intervention group)
  Neurofilament chains, light density (NfL)
Blood-based biomarkers of neuroplasticity | 4 weeks (Control group); 8 weeks (Intervention group)
  BDNF and GFAP. These will be measured using the same units of measurement

CONTACTS AND LOCATIONS:
Overall Officials: Lise B Worthen-Chaudhari, PhD, MFA, CMES, Principal Investigator — Ohio State University; Maryam B Lustberg, MD, MPH, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All data collected will be preserved and shared publicly upon publication to the NCI Cancer Research Data Commons (CRDC), a family of data repositories that provide cancer researchers with the ability to share diverse data types to maximize FAIR (i.e., Findable, Accessible, Interoperable, and Reusable) sharing of data. Shared data will be coded using unique filename identifiers that are not traceable to protected health information in order to enable future researchers to confirm results and/or incorporate these data in a metanalysis or similar larger study of relevant effects. The rationale is to share data for public access for other scientific learning and informational purposes to advance the knowledge base in these fields and to help researchers conduct secondary analysis on our broad range of datasets.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data will be made available upon publication within a peer-reviewed journal. Data will be available for as long as the NCI Cancer Research Data Commons (CRDC) supports access.
Access Criteria: Anyone with access to the NCI Cancer Research Data Commons (CRDC)

REFERENCES:
- [Background] Worthen-Chaudhari L, Bing J, Schmiedeler JP, Basso DM. A new look at an old problem: defining weight acceptance in human walking. Gait Posture. 2014;39(1):588-92. doi: 10.1016/j.gaitpost.2013.09.012. Epub 2013 Sep 28. PMID 24139684
- [Background] Worthen-Chaudhari L, Schnell PM, Hackney ME, Lustberg MB. Partnered dance evokes greater intrinsic motivation than home exercise as therapeutic activity for chemotherapy-induced deficits: secondary results of a randomized, controlled clinical trial. Front Psychol. 2024 Jun 19;15:1383143. doi: 10.3389/fpsyg.2024.1383143. eCollection 2024. PMID 38962217
- [Background] Worthen-Chaudhari LC, Crasta JE, Schnell PM, Lantis K, Martis J, Wilder J, Bland CR, Hackney ME, Lustberg MB. Neurologic dance training and home exercise improve motor-cognitive dual-task function similarly, but through potentially different mechanisms, among breast cancer survivors with chemotherapy-induced neuropathy: Initial results of a randomized, controlled clinical trial. J Alzheimers Dis. 2025 Jun;105(4):1114-1130. doi: 10.1177/13872877241291440. Epub 2024 Nov 25. PMID 39584292
- [Background] Worthen-Chaudhari L, Lamantia MT, Monfort SM, Mysiw W, Chaudhari AMW, Lustberg MB. Partnered, adapted argentine tango dance for cancer survivors: A feasibility study and pilot study of efficacy. Clin Biomech (Bristol). 2019 Dec;70:257-264. doi: 10.1016/j.clinbiomech.2019.08.010. Epub 2019 Aug 22. PMID 31751861
- [Background] Worthen-Chaudhari LC, Monfort SM, Bland C, Pan X, Chaudhari AMW. Characterizing within-subject variability in quantified measures of balance control: A cohort study. Gait Posture. 2018 Jul;64:141-146. doi: 10.1016/j.gaitpost.2018.05.031. Epub 2018 Jun 2. PMID 29908434
- [Background] Mezzanotte JN, Grimm M, Shinde NV, Nolan T, Worthen-Chaudhari L, Williams NO, Lustberg MB. Updates in the Treatment of Chemotherapy-Induced Peripheral Neuropathy. Curr Treat Options Oncol. 2022 Jan;23(1):29-42. doi: 10.1007/s11864-021-00926-0. Epub 2022 Feb 15. PMID 35167004
- [Derived] Luciani B, Carlson M, McNally G, Hackney ME, Crasta JE, Schnell P, Lustberg MB, Worthen-Chaudhari L. Dance-based avenues to advance nonpharmacologic treatment of chemotherapy effects (DAANCE): Study protocol for a multi-center, randomized controlled trial. Res Sq [Preprint]. 2025 Jul 7:rs.3.rs-6814353. doi: 10.21203/rs.3.rs-6814353/v1. PMID 40671809
- See also: The Jamesline — https://cancer.osu.edu